CLINICAL TRIAL: NCT07028723
Title: Relationship Between Proprioceptive Flexibility and the Occurrence of Lower Limb Ligament Injury in Pivot-contact Sports
Acronym: FlexiPro
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL25_0121; 2025-A00797-42 (Other: IdRCB)
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Lower Limb Ligament Injury
Keywords: Anterior Cruciate Ligament (ACL); Laterale Ankle Sprain (LAS); Inferior Tibio-fibular syndesmosis; Proprioception; Postural control; Injury Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- proprioceptive profile measurement (Experimental)
  Interventions: Other: proprioceptive profile measurement

INTERVENTIONS:
Other: proprioceptive profile measurement — Proprioceptive profile is measured by assessing static bipodal balance on a force platform. The patient is asked to stand motionless in bipodal support on a stable and then unstable floor, with vision masked by an eye mask. The investigators randomly apply a tendon vibration (80Hz) to the subjects' Achilles tendons or paravertebral muscles.
  This vibration alters proprioceptive information in the vibrated zone, leading to a disturbance in postural balance and an increased displacement of the center of pressure, whose position is continuously calculated from the force platform's sensors.
  Thus, depending on the amount of displacement of the center of pressure, the investigator calculates a proprioceptive weighting ratio (PWR) to deduce the weight assigned by the Central Nervous System to the various proprioceptive inputs during the postural task.
  An PWR of 1 indicates 100% use of information from the ankle, while an PWR of 0 means 100% use of information from the hip.

SUMMARY:
Among young athletes involved in pivot and pivot-contact sports (soccer, handball, rugby, etc.), lateral ankle sprains and lesions of the anterior cruciate ligament (ACL) are the most frequent ligament injuries. Despite existing prevention programs, these injuries lead to prolonged downtime, risk of recurrence and long-term sequelae.

A little-studied risk factor is proprioceptive rigidity, defined as the central nervous system's difficulty in adapting the use of sensory information (proprioception) according to environment and motor context. This deficit could limit the ability to maintain balance in high-risk situations, thereby increasing the likelihood of injury.

To our knowledge, there is no evidence of a direct link between proprioceptive profile (flexible/rigid) and the incidence of lower-limb ligament injury. If such a link is established, preventive strategies focusing on the recovery of an optimal proprioceptive profile could be developed in an attempt to limit the occurrence of ligament injuries in young elite and sub-elite athletes, and thus limit the medical, financial and personal repercussions for these athletes.

ELIGIBILITY:
Inclusion Criteria:

* Athlete practicing in a high-level program
* Aged between 14 and 25
* Practicing a pivot-contact sport (rugby, soccer, handball)

Exclusion Criteria:

* Lower limb injury <6 weeks prior to inclusion
* Concussion <6 weeks prior to inclusion
* Known neurological or vestibular disorder
* Lack of consent from athlete or legal guardians
* Non-affiliation with a social security scheme
* Persons under court protection
* Participant in another study with an ongoing exclusion period

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of occurrence of lower limb ligament injuries in groups of athletes with rigid proprioceptive profiles | During 1 year after inclusion
  Data collection on the occurrence of injuries will be carried out by club doctors, who will complete a questionnaire sent to them by e-mail by the investigator. They will then be contacted once a month by a single person to centralize the data.
Rate of occurrence of lower limb ligament injuries in groups of athletes with flexible proprioceptive profiles | During 1 year after inclusion
  Data collection on the occurrence of injuries will be carried out by club doctors, who will complete a questionnaire sent to them by e-mail by the investigator. They will then be contacted once a month by a single person to centralize the data.

SECONDARY OUTCOMES:
Describe the prevalence of rigid and flexible profiles in this population and according to the sport played (rugby, soccer, handball). | During 1 year after inclusion
Describe the relationship between proprioceptive stiffness and the period of training or match during which the injury occurred (training or match divided into 4) | During 1 year after inclusion
  Period of injury (1st, 2nd, 3rd or 4th quarter of training/match)
Describe the relationship between proprioceptive stiffness and the period of the season | During 1 year after inclusion
  Period of season (1st, 2nd, 3rd or 4th quarter of season)
Describe the relationship between proprioceptive stiffness and exposure time during training and matches | During 1 year after inclusion
  Number of hours of practice (training and match)
Describe the relationship between proprioceptive stiffness and injury mechanism (contact/non-contact) | During 1 year after inclusion
  Direct (contact) or indirect (non-contact) injury mechanism
Describe the relationship between proprioceptive stiffness and action during which injury occurs (attack/defense) | During 1 year after inclusion
  Action of injury (attack or defense)
Describe the relationship between proprioceptive stiffness and occurrence of a first or recurrent injury | During 1 year after inclusion
  First episode or recurrence
Describe the relationship between proprioceptive stiffness and time to return to sport at the same level | During 1 year after inclusion
  Time to return to sport at same level

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided